CLINICAL TRIAL: NCT00574691
Title: ECLIPSE Feasibility Trial (Ensure's Vascular Closure Device Speeds Hemostasis) Trial
Brief Title: ECLIPSE Feasibility Trial (Ensure's Vascular Closure Device Speeds Hemostasis Trial) EU
Acronym: ECLIPSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll - Director Clinical Affairs, Cordis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM 06-01EU
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary; Coronary Arteriosclerosis
Keywords: Closure Device; Angiography; Angioplasty; Hemostasis; Heart Catheterization; Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Vascular Closure Device
  Interventions: Device: 7F Ensure Medical Vascular Closure Device

INTERVENTIONS:
Device: 7F Ensure Medical Vascular Closure Device — Vascular Closure Device
  Other Names: Ensure Medical Vascular Closure Device

SUMMARY:
To assess the safety and feasibility of the 7F Ensure Medical Vascular Closure Devices to facilitate hemostasis in patients undergoing diagnostic or interventional procedures.

DETAILED DESCRIPTION:
Multi-center (up to 6 European sites), non-blinded, non-randomized, feasibility study with a 2-month enrollment period and 30-day clinical follow-up.

60 patients (plus up to 36 "roll-in" device training patients) undergoing diagnostic or interventional coronary or peripheral procedures utilizing a 7F arterial puncture in the common femoral artery. Patients are excluded if they have a previous target artery closure with any closure device, recent myocardial infarction or thrombolytic therapy, treatment with thrombin-specific anticoagulants or low molecular weight heparin, fluoroscopically visible calcium or atherosclerosis ≤ 1 cm of puncture site, or planned target site access ≤ 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 85 years of age
* Patient/legal representative provides written informed consent
* Patient is scheduled for a coronary or peripheral diagnostic or interventional procedure
* Patient is able to undergo emergent vascular surgery if a complication related to the VCD necessitates such surgery
* Patient has a 7F arterial puncture located in the common femoral artery
* Target vessel has a lumen diameter ≥ 5 mm
* Patient is willing and able to complete follow-up
* Catheterization procedure is planned and elective

Exclusion Criteria:

* Arterial puncture in the femoral artery of both legs
* Prior target artery closure with any closure device or closure with manual compression ≤ 30 days prior to the cardiac or peripheral catheterization procedure
* Patients with a history of significant bleeding or with any known or documented bleeding disorders, such as Thrombocytopenia (with < 100,000 platelet count), Von Willebrand's disease, anemia (Hgb < 10 g/dL, Hct < 30%), thrombasthenia, decreased fibrinogen (< 200 mg/dL), and Factor V deficiency
* Acute ST-elevation myocardial infarction ≤ 48 hours prior to the cardiac or peripheral catheterization procedure
* Uncontrolled hypertension (BP ≥ 180/110 mmHg)
* Heparinized patients with elevated pre-closure ACT level:> 250 seconds with GP IIb/IIIa inhibitor > 300 seconds no GP IIb/IIIa inhibitor
* Patient is ineligible for in-lab catheterization lab introducer sheath removal
* Concurrent participation in another investigational device or drug trial
* Thrombolytic therapy (e.g. streptokinase, urokinase, t-PA) ≤ 24 hours prior to the cardiac or peripheral catheterization procedure
* Angiomax (bivalirudin) or other thrombin-specific anticoagulants or low molecular weight heparin ≤ 24 hours prior to the cardiac or peripheral catheterization procedure
* Evidence of a preexisting hematoma, arteriovenous fistula, or pseudoaneurysm at the access site prior to start of femoral artery closure procedure
* Prior femoral vascular surgery or vascular graft in region of access site or contralateral common femoral artery
* The targeted femoral artery is tortuous or requires an introducer sheath length > 11 cm
* Fluoroscopically visible calcium, atherosclerotic disease, or stent ≤ 1 cm of the puncture site that would interfere with the placement of the VCD's plug
* Difficulty in obtaining vascular access resulting in multiple arterial punctures and/or posterior arterial puncture
* Antegrade puncture
* BMI > 40 kg/m2
* Symptomatic leg ischemia in the target vessel limb including severe claudication (< 50 meter) or weak/absent pulse
* Targeted femoral artery diameter stenosis ≥ 50%
* Pre-existing severe non-cardiac systemic disease or pre-existing terminal illness
* Planned arterial access at the same access site ≤ 30 days following the femoral artery closure procedure
* Patient has known allergy to any materials used in the VCD
* Patient is known to require an extended hospitalization (e.g. patient is undergoing CABG surgery)
* Pre-existing systemic or cutaneous infection
* Prior or recent use of an intra-aortic balloon pump through the arterial access site
* Cardiogenic shock (hemodynamic instability requiring intravenous medications or mechanical support) experienced during or immediately post-catheterization
* Patient is unable to ambulate at baseline
* Patient is known or suspected to be pregnant, or is lactating
* Patient has already participated in this trial
* Patient has known allergy to contrast medium
* Patient is unavailable for follow-up
* Any angiographic or clinical evidence that the investigator feels would place the patient at increased risk with the use of the VCD
* Required simultaneous ipsilateral or contralateral venous puncture

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2007-06; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Time to hemostasis and time to ambulation. | at time introducer sheath is removed
Combined rate of the following SAEs:Vascular injury or repair; access site bleeding, infection, nerve injury; ipsilateral lower extremity ischemia. | 30 days

SECONDARY OUTCOMES:
Device success. | initial hemostasis time ≤ 5 minutes and removal of the intact delivery system
Procedural success. | 30 days
Time the patient is deemed eligible for hospital discharge. | time of the access site closure until patient is discharge
Rebleeding following initial hemostasis requiring a subsequent intervention. | prior to hospital discharge, and at the 30-day follow-up
Pseudoaneurysm not requiring treatment. | prior to hospital discharge, and at the 30-day follow-up
Pseudoaneurysm treated with ultrasound-guided thrombin injection or ultrasound-guided fibrin adhesive injection. | prior to hospital discharge, and at the 30-day follow-up
Arteriovenous fistula documented by ultrasound or CT scan. | prior to hospital discharge, and at the 30-day follow-up
Access site hematoma ≥ 6 cm. | prior to hospital discharge, and at the 30-day follow-up
Post-hospital discharge access site-related bleeding. | prior to hospital discharge, and at the 30-day follow-up
Access site-related bleeding requiring > 30 minutes to achieve hemostasis. | prior to hospital discharge, and at the 30-day follow-up
Ipsilateral lower extremity arterial emboli. | prior to hospital discharge, and at the 30-day follow-up
Transient loss of ipsilateral lower extremity pulse. | prior to hospital discharge, and at the 30-day follow-up
Ipsilateral deep vein thrombosis. | prior to hospital discharge, and at the 30-day follow-up
Access site-related vessel laceration. | prior to hospital discharge, and at the 30-day follow-up
Transient access site-related nerve injury | prior to hospital discharge, and at the 30-day follow-up
Access site wound dehiscence. | prior to hospital discharge, and at the 30-day follow-up
Localized access site infection treated with oral antibiotics. | prior to hospital discharge, and at the 30-day follow-up
Retroperitoneal bleeding. | prior to hospital discharge, and at the 30-day follow-up
Ipsilateral peripheral artery total occlusion. | prior to hospital discharge, and at the 30-day follow-up
Ecchymosis ≥ 6 cm. | prior to hospital discharge, and at the 30-day follow-up
Intraluminal plug delivery not requiring surgical intervention. | prior to hospital discharge, and at the 30-day follow-up
Decrease in pedal pulse. | prior to hospital discharge, and at the 30-day follow-up
Death. | prior to hospital discharge, and at the 30-day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Wiemer, Dr., Principal Investigator — Herz-und Diabeteszentrum NRW
Locations (1):
- Herz-und Diabeteszentrum NRW, Bad Oeynhausen, Germany

REFERENCES:
- [Derived] Wiemer M, Langer C, Fichtlscherer S, Firschke C, Hofbauer F, Lins M, Haude M, Debefve C, Stoll HP, Hanefeld C. First-in-man experience with a new 7F vascular closure device (EXOSEAL): the 7F ECLIPSE study. J Interv Cardiol. 2012 Oct;25(5):518-25. doi: 10.1111/j.1540-8183.2012.00739.x. Epub 2012 Jul 5. PMID 22762417